CLINICAL TRIAL: NCT06129110
Title: Effect of Weight Loss on Intermuscular Adipose Tissue (IMAT) Signaling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 23-0545; 1R01DK134706-01A1 (NIH)
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Insulin Sensitivity; Muscle Weakness; Adiposity; Insulin Resistance
Keywords: IMAT; Intermuscular Adipose Tissue; Weight Loss; Diet
MeSH Terms: conditions — Obesity; Insulin Resistance; Muscle Weakness; Weight Loss | interventions — Diet, Reducing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet Weight Loss (Experimental): Low calorie meal replacement shakes
  Interventions: Behavioral: Diet Weight Loss
- Delayed Intervention (No Intervention): Normal feeding

INTERVENTIONS:
Behavioral: Diet Weight Loss — Low calorie diet of meal replacement shakes
  Arms: Diet Weight Loss

SUMMARY:
The goal of this intervention study is to learn about how weight loss impacts molecular signaling of intermuscular adipose tissue (IMAT) in individuals with obesity. The main question it aims to answer is how inflammatory molecules secreted by IMAT promote muscle insulin resistance and inflammation, and how these same molecules are diminished after weight loss. Following screening visits involving body composition measures, blood testing, strength testing, and a thigh muscle biopsy, participants will go through a 12-week dietary intervention for weight loss. After 12 weeks, this will be followed by the same testing and biopsies that were completed before the intervention. Researchers will then compare outcomes of individuals who lost weight to individuals who did not lose weight.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy men and women aged 18-70
* BMI between 30-40
* Less than 1 hour of exercise per week
* Women:

  1. may be pre or post menopausal

Exclusion Criteria:

* Type 1 or Type 2 diabetes
* Thyroid disease
* History of lung disease
* Active use of nicotine
* Severe plasma lipid disorders
* Taking hormone replacement drugs, blood thinners, or thiazoladinediones
* Women:

  1. Currently going through menopause or peri-menopause
  2. Pregnant or breastfeeding
  3. History of Polycystic Ovary Syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Insulin Sensitivity | 12 weeks
  Participants will undergo a standard 3-hour hyperinsulinemic/euglycemic clamp with insulin infused at 80 mU/m2/min, and glucose clamped at 90 mg/dl with a variable dextrose infusion.
Body Weight | 12 weeks
  Participant weight will be measured using BodyTrace scales during the 12 week intervention.
IMAT Content | 12 weeks
  A multi-slice MRI will be used to quantify IMAT and muscle content in both legs with acquisition of ~20 axial images (10 mm thickness) with 10 mm spacing between images starting superior to the patella. IMAT content will be quantified using the well-validated Sirlin 6-echo method and normalized to muscle volume.
Muscle Mass | 12 weeks
  A multi-slice MRI will be used to quantify IMAT and muscle content in both legs with acquisition of ~20 axial images (10 mm thickness) with 10 mm spacing between images starting superior to the patella. Muscle volume will be quantified using standard methods with anatomical cross-sectional area evaluated in each T1 weighted, high resolution, gradient echo profile scan, and multiplied by the length of the muscle.
Muscle Strength | 12 weeks
  Participants will perform quadriceps muscle strength testing using an isokinetic dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No